CLINICAL TRIAL: NCT06010602
Title: COMPARISON OF THE POSTOPERATIVE ANALGESIC EFFECTIVENESS OF QUADRATUS LUMBORUM BLOCK and ILIOINGUINAL -ILIOHIPOGASTRIC NERVE BLOCK IN CESAREAN SECTION OPERATIONS
Brief Title: Postoperative Analgesia in Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GaziosmanpasaTREH47
Record Dates: First submitted 2023-08-20; First posted 2023-08-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Pain
Keywords: cesarean section; Quadratus lumborum III block; Ilioinguinal iliohypogastric block; analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus lumborum block group (Active Comparator): the patient In the lateral decubitus position, a subcostal area and above the iliac crest in the mid-axillary line, a convex ultrasound probe is placed under sterile conditions. Using an in-plane technique, the quadratus lumborum and psoas major muscles, as well as the transverse process of the L4 vertebra, are visualized. 22G, 100 mm peripheral block needle is used to perform the block. The needle is directed between the quadratus lumborum muscle and the psoas major muscle in the subfascial plane, following hydrodissection for proper needle placement. Then, 20 mL of 0.25% bupivacaine is injected slowly, aspirating every 5 cc to ensure proper spread. The injection is performed under ultrasound guidance, visualizing the local anesthetic pushing the fascia. The same procedure will be repeated for the other side.
  Interventions: Procedure: Quadratus lumborum block
- İlioinguinal-İliohipogastric nerve block group (Active Comparator): the patient in the supine position, a linear ultrasound probe is placed over the spina iliaca anterior superior (SIAS) line, drawn from SIAS to the umbilicus. The probe is used to visualize the abdominal wall muscles, focusing on the fascial plane between the transversus abdominis and internal oblique muscles, where a flattened football-like appearance is seen. The iliohypogastric nerve is observed more laterally, and the ilioinguinal nerve is seen more medially. Using an in-plane technique with 22G, 100 mm peripheral block needle, local anesthetic is injected near the SIAS, between the transversus abdominis and internal oblique muscles. Again, 20 mL of 0.25% bupivacaine is injected slowly, aspirating every 5 cc, and the injection is visualized under ultrasound guidance, ensuring proper fascial spread. The same procedure will be repeated for the other side.
  Interventions: Procedure: İlioinguinal-İliohipogastric nerve block

INTERVENTIONS:
Procedure: Quadratus lumborum block — For all patients, postoperative analgesia was planned as paracetamol 1g four times a day for the first 24 hours after surgery. Patients with Numeric Rating Scale (NRS) scores greater than 3 at 2, 4, 8, 12, and 24 hours postoperatively were administered rescue analgesia with tramadol hydrochloride at a dose of 1mg/kg.
  Other Names: Intravenous analgesic medication
  Arms: Quadratus lumborum block group
Procedure: İlioinguinal-İliohipogastric nerve block — For all patients, postoperative analgesia was planned as paracetamol 1g four times a day for the first 24 hours after surgery. Patients with Numeric Rating Scale (NRS) scores greater than 3 at 2, 4, 8, 12, and 24 hours postoperatively were administered rescue analgesia with tramadol hydrochloride at a dose of 1mg/kg.
  Other Names: Intravenous analgesic medication
  Arms: İlioinguinal-İliohipogastric nerve block group

SUMMARY:
İn this study, planned to compare the post-operative analgesic efficacy of Ilioinguinal iliohypogastric (II-IH) nerve block and Quadratus lumborum III Block in elective cesarean section operations.

this study primary aim is; To compare and evaluate the first rescue analgesia requirement times after Quadratus lumborum III and II-IH Block for postoperative analgesia after elective cesarean section operations under spinal anesthesia.

Our secondary aims are:

1. To compare the amount of total analgesic use in the first 24 hours in patients
2. To compare the NRS (Numering rating scale) values (resting and dynamic) at 2. 4. 8. 12 . 24. hours in the postoperative follow-up of the patients
3. Comparing the side effects such as postoperative nausea and vomiting

DETAILED DESCRIPTION:
Patients who underwent elective cesarean section under spinal anesthesia will be divided into two groups at the end of the operation, using the closed envelope randomization method as Quadratus lumborum III and II-IH nerve block. Spinal anesthesia will be applied to all patients who will undergo elective cesarean section. At the end of the operation, they will be taken to the postoperative block room. All blocks will be performed by the same anesthesiologist under USG guidance. 20 ml of 0.25% bupivacaine will be used in the blocks. All patients will be followed in the block room for 30 minutes after the block application. Patients with a Modified Aldret score above 8 will be sent to the service because they are under spinal anesthesia at the end of the operation.At the end of the operation, when the spinal level regresses to two dermatome levels, paracetamol 1gr IV will be administered to all patients for post-op analgesia.Postoperative analgesia was planned for the patients as paracetamol 4x1 gr. Tramadol hydrochloride 1mg/kg was planned as rescue analgesia in the ward for patients with NRS scores greater than 3 in their postoperative follow-up.

Patients 2.,4.,8.,12.,24. hours will be followed by an anesthesia assistant who is different from the researcher who applied the block and who is blind for the study. The patients' first rescue analgesia times, NRS scores, postoperative side effects, and total analgesic amounts used in 24 hours will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 40
* ASA 2 risk group
* Patients at 37-41 weeks of pregnancy
* undergoing cesarean section under spinal anesthesia

Exclusion Criteria:

* The patient does not accept the procedure.
* Patients with a history of eclampsia and preeclampsia during pregnancy
* local anesthetic allergy
* Infection at the procedure site
* Anticoagulant use with bleeding disorder
* Chronic analgesia and opioid use
* Mental, psychiatric and neurological problems
* Patients with ASA 3 and above with a history of any chronic disease.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Comparison of first rescue analgesia | 24 hour
  For all patients, postoperative analgesia was planned as paracetamol 1g four times a day for the first 24 hours after surgery. Patients with Numeric Rating Scale (NRS) scores greater than 3 at 2, 4, 8, 12, and 24 hours postoperatively will receive rescue analgesia with tramadol hydrochloride at a dose of 1mg/kg. The time of the first administration of tramadol hydrochloride for each patient will be compared.

SECONDARY OUTCOMES:
comparing the amount of total analgesic use in the first 24 hours in patients | 24 hours
  For all patients, postoperative analgesia was planned as paracetamol 1g four times a day for the first 24 hours after surgery. Patients with Numeric Rating Scale (NRS) scores greater than 3 at 2, 4, 8, 12, and 24 hours postoperatively will receive rescue analgesia with tramadol hydrochloride at a dose of 1mg/kg.The total tramadol consumption of patients within the first 24 hours will be compared.
Comparing the NRS values in 2,4,8,12,24 hours in the postoperative follow-up of the patients | 24 hours
  To compare the Numeric Rating Scale (NRS) values (at rest and with movement) of the patients during postoperative follow-ups at 2, 4, 8, 12, and 24 hours.
Comparing side effects such as postoperative nausea and vomiting | 24 hours
  To compare postoperative side effects such as nausea and vomiting within the first 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: serpil sehirlioglu, Principal Investigator — Gaziosmanpasa Research and Education Hospital
Locations (1):
- Gaziosmanpasa Research and Education Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Irwin R, Stanescu S, Buzaianu C, Rademan M, Roddy J, Gormley C, Tan T. Quadratus lumborum block for analgesia after caesarean section: a randomised controlled trial. Anaesthesia. 2020 Jan;75(1):89-95. doi: 10.1111/anae.14852. Epub 2019 Sep 15. PMID 31523801
- [Result] Yetik F, Yilmaz C, Karasu D, Haliloglu Dastan N, Dayioglu M, Baytar C. Comparison of ultrasound-guided quadratus lumborum block-2 and quadratus lumborum block-3 for postoperative pain in cesarean section: A randomized clinical trial. Medicine (Baltimore). 2022 Dec 9;101(49):e31844. doi: 10.1097/MD.0000000000031844. PMID 36626453
- [Result] Koksal E, Aygun H, Genc C, Kaya C, Dost B. Comparison of the analgesic effects of two quadratus lumborum blocks (QLBs), QLB type II vs QLB type III, in caesarean delivery: A randomised study. Int J Clin Pract. 2021 Oct;75(10):e14513. doi: 10.1111/ijcp.14513. Epub 2021 Jun 23. PMID 34117829
- [Result] Staker JJ, Liu D, Church R, Carlson DJ, Panahkhahi M, Lim A, LeCong T. A triple-blind, placebo-controlled randomised trial of the ilioinguinal-transversus abdominis plane (I-TAP) nerve block for elective caesarean section. Anaesthesia. 2018 May;73(5):594-602. doi: 10.1111/anae.14222. Epub 2018 Jan 29. PMID 29377066